CLINICAL TRIAL: NCT02547337
Title: Glucose-stimulated Pancreatic Islet and Intestinal Blood Flow in Healthy Subjects and in Type 1 Diabetes Using Positron Emission Tomography and Diffusion Weighted Imaging
Brief Title: Glucose-stimulated Pancreatic Islet and Intestinal Blood Flow in Healthy Subjects and in Type 1 Diabetes
Acronym: ISLET-PET
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Pirjo Nuutila, MD, Prof., Turku University Hospital
Other Study IDs: ISLET-PET
Record Dates: First submitted 2015-09-02; First posted 2015-09-11 (Estimated); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, serum, faeces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 diabetes
- Healthy subjects

SUMMARY:
Type 1 diabetes is the major type of diabetes in the young. The pathophysiology still needs clarification in order to reach feasible means of preventing the disease. This study aims in defining the differences in pancreatic and intestinal blood flow between subjects with and without type 1 diabetes and validating the methodology to achieve this. Earlier animal studies have demonstrated changes in pancreatic islet blood flow using microspheres. The aim of this study is to test and validate a method for the assessment of islet perfusion in humans using molecular imaging. The investigators hypothesize that glucose-stimulated pancreatic perfusion is enhanced specifically in islets in healthy subjects and that this increase is mostly suppressed in subjects with type 1 diabetes.

Positron emission tomography (PET) is a non-invasive imaging technique, which can be used to study flow and metabolism of different organs. Using radiowater ([15O]H2O) and PET, cellular perfusion can be measured directly and noninvasively. Recently, diffusion weighted magnetic resonance imaging (DWI) has also been applied as a complimentary method for the assessment to quantitate changes in pancreatic blood flow.

In the study 10 healthy subjects and 10 subjects with type 1 diabetes will be imaged on two separate days. Pancreatic and intestinal perfusion are first measured with [15O]H2O and combined PET/magnetic resonance imaging before and 5 and 15 minutes after intravenous glucose infusion. On the second day, PET imaging is replaced by dynamic DWI conducted in the same time schedule and with intravenous glucose stimulation.

ELIGIBILITY:
Criteria for healthy subjects

Inclusion criteria

* Healthy as judged by history and examination
* Age 18-30 years
* Body mass index (BMI) 18 - 27 kg/m2
* Normal 2 h oral glucose tolerance test

Exclusion criteria

* Any chronic disease
* Pregnancy
* Blood pressure > 140/90 mmHg
* Smoking
* Presence of any ferromagnetic objects in the body
* Any other condition that could possibly create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of the study results

Criteria for subjects with type 1 diabetes (T1D)

Inclusion criteria

* T1D diagnosed at least 5 years ago
* Age 18-30 years
* BMI 18 - 30 kg/m2
* Good or moderate glycemic control with long-acting insulin analogue combined with injections of rapid-acting insulin
* Uncomplicated T1D or with minor microvascular complications

Exclusion criteria

* Any other condition or disease possibly affecting circulation, as evaluated by a physician
* Pregnancy
* Blood pressure > 140/90 mmHg
* Smoking
* Presence of any ferromagnetic objects in the body
* Any other condition that could possibly create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of the study results

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects recruited via newspaper advertisements. Subjects with Type 1 diabetes recruited at the policlinics of endocrinology and internal medicine in the district of Turku University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Pancreatic islet blood flow acquired with PET and DWI (ml ml-1 min-1) | within one study day
  healthy subjects and subjects with T1DM are studied once using imaging
Intestinal blood flow acquired with PET and DWI (ml ml-1 min-1) | within one study day
  healthy subjects and subjects with T1DM are studied once using imaging

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, Prof., Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland